CLINICAL TRIAL: NCT03894865
Title: Screening and Prevalence of Adolescent Idiopathic Scoliosis in Selected Urban and Countryside Schools in Egypt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima Abdelaty Hassan, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: scoliosis in Egypt
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Scoliosis
Keywords: scoliosis, prevalence; screening, Egypt
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- urban school (Experimental): Male students from selected urban schools undergo screening for idiopathic scoliosis
  Interventions: Other: procedure1; Other: procedure2
- countryside schools (Experimental): Male students from selected countryside schools undergo screening for idiopathic scoliosis
  Interventions: Other: procedure1; Other: procedure2

INTERVENTIONS:
Other: procedure1 — The students will be asked to bend forward with his knees straight, feet together and hands freely and loosely hanged. if there was scoliosis the rib cage rotated and a hump appeared. Positive test indicated the presence of a rib hump and negative if there was any hump appeared
  Other Names: Adam's forward bend test
Other: procedure2 — Measurement of the angle of trunk rotation (ATR) by using a scoliometer HD smartphone application.
  Other Names: Angle of trunk rotation

SUMMARY:
Early detection of scoliosis and determination of which areas are more affected urban or countryside will help in early management. Also, this will guide the government and the community for early intervention to decrease the factors that leads to this postural abnormality. This also will guide another clinician to search for the cause of these posture deformities and to concentrate screening for special areas with special cultures.

DETAILED DESCRIPTION:
Scoliosis may have an impact on the Egyptian society as children between 10-15 years old represent 9.5 % of the population which is the third large category appendix (3). So without the early detection of adolescent idiopathic scoliosis for that age group, bad impacts will be implemented for Egyptian society by causing disabilities and psychological problems for these children.

The early detection of scoliosis is of a great importance as curve detection before skeletal maturation gives a good opportunity for early treatment or prevention of curve progression. Scoliosis has a bad effect on cosmetic appearance, quality of life, Psychological well-being, disability, back Pain, breathing function. It may also progress in adulthood and need further treatment. So a multidimensional and comprehensive evaluation of scoliosis patients is necessary to design a complete therapeutic approach.

ELIGIBILITY:
Inclusion criteria:

1. Age range from 10 to 15 years.
2. Males students.
3. Students who have structural scoliosis.

Exclusion criteria:

1. Congenital deformities.
2. Recent fracture and there is a fixation in the upper or the lower extremities
3. Neuromuscular disorder (Cerebral palsy and spinal muscle atrophy).
4. Syndromic disorders (Muscular dystrophy, Osteogenesis imperfect, and Spina-bifida).

Ages: 10 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 840 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Positive Adam's forward bending test | 10 minutes
  Proportion of patients with a positive Adam's forward bending test
degree of trunk rotation | 15 minutes
  scoliometer HD reading >7 degrees (=>20 degrees Cobb angle) Proportion of patients with more than 7 degree

SECONDARY OUTCOMES:
screening | 15 minutes
  percentage of childerns with idiopathic scoliosis

CONTACTS AND LOCATIONS:
Overall Officials: karima A Hassan, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No